CLINICAL TRIAL: NCT04562766
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo Controlled, Parallel-Group Study With an Open-Label Extension to Evaluate the Efficacy and Safety of Oral Rilzabrutinib (PRN1008) in Adults and Adolescents With Persistent or Chronic Immune Thrombocytopenia (ITP)
Brief Title: Study to Evaluate Rilzabrutinib in Adults and Adolescents With Persistent or Chronic Immune Thrombocytopenia (ITP)
Acronym: LUNA 3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Principia Biopharma, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC17093; PRN1008-018 (Other: Sanofi Identifier); 2023-509401-71 (Registry Identifier: CTIS)
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rilzabrutinib (Experimental): Patients receive rilzabrutinib 400mg orally twice daily for up to 24 weeks followed by 28 weeks of open label period
  Interventions: Drug: Rilzabrutinib
- Placebo (Placebo Comparator): Patients receive matching placebo 400mg orally twice daily for up to 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rilzabrutinib — 400mg Caplet
  Other Names: PRN1008
  Arms: Rilzabrutinib
Drug: Placebo — 400mg Caplet
  Other Names: PRN1008 Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind study of rilzabrutinib in patients with persistent or chronic ITP, with an average platelet count of <30,000/μL (and no single platelet count >35,000/μL) on two counts at least 5 days apart in the 14 days before treatment begins. Patients will receive rilzabrutinib or placebo 400mg twice daily.

For each patient, the study will last up to 60 weeks from the start of the Screening Period to the End of Study (EOS) visit. This includes Screening (up to 4 weeks) through a 12 to 24-week Blinded Treatment Period followed by a 28-week Open-Label Period. Followed by a 4-week post dose follow-up.

For adult participants, the maximum duration of the long-term extension (LTE) period will be 12 months from the date of the last adult participant to enter the LTE.

For pediatric participants, the maximum duration of the LTE period will be 12 months from the date of the last pediatric participant to enter the LTE.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will be male and female with primary ITP with duration of >6 months in pediatric participants aged 12 to <18 years (pediatric participants aged 10 to <12 years will be enrolled in the EU [EEA countries] only) and duration of >3 months in ages 18 years and above
2. Patients who had a response (achievement of platelet count ≥50,000/µL) to IVIg/anti-D or CSs that was not sustained and who have documented intolerance, insufficient response or any contra-indication to any appropriate courses of standard of care ITP therapy
3. An average of 2 platelet counts at least 5 days apart of <30,000/µL during the Screening period and no single platelet count >35,000/µL, within 14 days prior to the first dose of study drug.

   - Pediatric patients must additionally be determined to need treatment for ITP as per clinical assessment by the Investigator.
4. Adequate hematologic, hepatic, and renal function (absolute neutrophil count ≥1.5 X 10^9/L, AST/ALT ≤1.5 x upper limit of normal [ULN], albumin ≥3 g/dL, total bilirubin ≤1.5 x ULN [unless the patient has documented Gilbert syndrome], glomerular filtration rate >50 [Cockcroft and Gault method for adult and Bedside Schwartz Equation for Pediatric participants])
5. Hemoglobin >9 g/dL within 1 week prior to Study Day 1
6. All contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies
7. Patients must be able to provide written informed consent or informed assent with corresponding informed consent obtained from the patient's guardian and agree to the schedule of assessments

Exclusion Criteria:

1. Patients with secondary ITP
2. Pregnant or lactating women
3. History (within 5 years of Study Day 1) or current, active malignancy requiring or likely to require chemotherapeutic or surgical treatment during the study, with the exception of non melanoma skin cancer
4. Transfusion with blood, blood products, plasmapheresis, or use of any other rescue medications with intent to increase platelet count within 14 days before Study Day 1
5. Change in CS and/or TPO-RA dose within 14 days prior to Study Day 1 (more than 10% variation from current doses)
6. Immunosuppressant drugs other than CSs within 5 times the elimination half-life of the drug or 14 days of Study Day 1, whichever is longer
7. Treatment with rituximab or splenectomy within the 3 months prior to Study Day 1

   - Patients treated with rituximab will have normal B-cell counts prior to enrollment
8. Has received any investigational drug within the 30 days before receiving the first dose of study medication, or at least 5 times elimination half-life of the drug (whichever is longer); patient should not be using an investigational device at the time of dosing

   * Patients who previously received treatment with Bruton's Tyrosine Kinase (BTK) inhibitors (except rilzabrutinib) within 30 days before the first dose of study drug are not eligible
   * Patients who previously received rilzabrutinib at any time are not eligible
9. History of solid organ transplant
10. Myelodysplastic syndrome
11. Live vaccine within 28 days prior to Study Day 1 or plan to receive one during the study
12. Planned surgery in the time frame of the dosing period

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2026-08-26 (Estimated)

PRIMARY OUTCOMES:
Durable platelet response during the last 6 weeks of the 24-week blinded treatment period (not for EU and UK) | 24 weeks
  Durable platelet response is defined as a proportion of participants able to achieve platelet counts at or above 50,000/μL for ≥ two-thirds of at least 8 non-missing weekly scheduled platelet measurements during the last 12 weeks of the 24-week blinded treatment period in the absence of rescue therapy, provided that at least 2 non-missing weekly scheduled platelet measurements are at or above 50,000/μL.
for EU and UK: Proportion of adult participants able to achieve platelet counts at or above 50,000/μL for at least 8 out of the last 12 weeks of the 24-week blinded treatment period in the absence of rescue therapy | 24 weeks

SECONDARY OUTCOMES:
Number of weeks with platelet count ≥50,000/μL OR between ≥30,000/μL and <50,000/μL and at least doubled from baseline over the 24-week blinded treatment period in the absence of rescue therapy | 24 weeks
Number of weeks with platelet counts ≥30,000/μL and at least doubled from baseline over the 24-week blinded treatment period in the absence of rescue therapy | 24 weeks
Time to first platelet count of ≥50,000/μL OR between ≥30,000/μL and <50,000/μL and doubled from baseline | 24 weeks
Proportion of patients requiring rescue therapy during the 24-week blinded treatment period | 24 weeks
Change from baseline on Item 10 of the ITP-Patient Assessment Questionnaire in adult patients (≥18 years) at Week 13 | From baseline to Week 13
for EU and UK: Change from baseline in Idiopathic Thrombocytopenic Purpura Bleeding Scale (IBLS) assessment at Week 25 | At Week 25
Proportion of participants who able to achieve stable platelet response, within a period of 24 weeks following initial achievement of the platelet response | 24 weeks
  Stable platelet response is defined as no 2 scheduled visits, at least 4 weeks apart, with a platelet count less than 50,000/µL, without an intervening visit with a platelet count ≥50,000/µL. Initial platelet response defined as platelet count ≥50,000/μL within 12 weeks of initiation of treatment with rilzabrutinib during the study.
Frequency and severity of Treatment Emergent Adverse Events | 52 weeks of treatment, 12 months of long term extension and 4 weeks of follow up post last dose
  Including physical examination, ECG, clinical laboratory test results, vital signs and laboratory tests (serum chemistry, hematology, except for platelet counts included in the primary efficacy endpoint)
Frequency and severity of bleeding TEAEs | 52 weeks of treatment, 12 months of long term extension and 4 weeks of follow up post last dose
Plasma concentrations of rilzabrutinib | Until 52 weeks
Change from baseline on the Symptoms, Bother and Activity domains of the ITP Patient Assessment Questionnaire (ITP-PAQ) in adult patients (≥18 years) | 52 weeks of treatment, 12 months of long term extension and 4 weeks of follow up post last dose
  The ITP Patient Assessment Questionnaire™ (ITP-PAQ™) is a disease-specific instrument that was designed to measure the Quality of Life (QoL) of adult patients with immune thrombocytopenia. The items employ a 4-week recall with responses recorded on 4-, 5- or 7-point Likert scales. All item scores are transformed to a 0 to 100 continuum where higher scores represent better QoL and are weighted equally to derive the scale scores.
Change from baseline in disease-specific QoL as measured by the Kids' ITP Tools (ITP-KIT) score in pediatric participants | 52 weeks of treatment, 12 months of long term extension and 4 weeks of follow up post last dose
  The ITP-KIT include a battery of three disease-specific instruments, a child self-report form designed to be completed by children ≥7 years, a parent proxy report form for children <7 and a parent impact form. Respondents record their disease experience based on a 1-week recall. The instrument yields a total score which is the summation of the items converted to a 0 to 100 score with higher scores indicating better disease-specific QoL.

CONTACTS AND LOCATIONS:
Locations (155):
- United States (17):
  - University of Southern California_Investigational Site Number 84024, Los Angeles, California
  - UCSF Benioff Children's Hospital San Francisco_Investigational Site Number 84020, San Francisco, California
  - Lundquist Institute for Biomedical Innovation at Harbor UCLA Medical Center_Investigational Site Number 84037, Torrance, California
  - The Oncology Institute of Hope and Innovation_Investigational Site Number 84031, Whittier, California
  - Children's Hospital Colorado_Investigational Site Number 84025, Aurora, Colorado
  - IMMUNOe International Research Centers_Investigational Site Number 84028, Centennial, Colorado
  - ASCLEPES Research Centers_Investigational Site Number 84023, Weeki Wachee, Florida
  - Children's Healthcare of Atlanta_Investigational Site Number 84034, Atlanta, Georgia
  - Rush University Medical Center_Investigational Site Number 84029, Chicago, Illinois
  - University of Louisville - James Graham Brown Cancer Center_Investigational Site Number 84033, Louisville, Kentucky
  - Massachusetts General Hospital Site Number : 84038, Boston, Massachusetts
  - Montefiore Medical Center_Investigational Site Number 84032, The Bronx, New York
  - University Hospitals Cleveland Medical Center Site Number : 84036, Cleveland, Ohio
  - Cleveland Clinic_Investigational Site Number 84026, Cleveland, Ohio
  - The Children's Hospital of Philadelphia (CHOP)_Investigational Site Number 84027, Philadelphia, Pennsylvania
  - University of Utah-Huntsman Cancer Institute_Investigational Site Number 84035, Salt Lake City, Utah
  - University of Washington Medical Centre Site Number : 84041, Seattle, Washington
- Argentina (5):
  - Investigational Site Number : 3206, Capital Federal, Buenos Aires
  - Investigational Site Number : 3211, La Plata, Buenos Aires
  - Investigational Site Number : 3205, Córdoba, Córdoba Province
  - Investigational Site Number : 3209, Corrientes
  - Investigational Site Number : 3208, San Juan
- Australia (6):
  - Investigational Site Number : 3607, Kogarah, New South Wales
  - Investigational Site Number : 3608, Westmead, New South Wales
  - Investigational Site Number : 3611, Brisbane, Queensland
  - Investigational Site Number : 3609, Adelaide, South Australia
  - Investigational Site Number : 3606, Frankston, Victoria
  - Investigational Site Number : 3610, Perth, Western Australia
- Austria (5):
  - Investigational Site Number : 4005, Graz
  - Investigational Site Number : 4004, Leoben
  - Investigational Site Number : 4001, Linz
  - Investigational Site Number : 4003, Steyr
  - Investigational Site Number : 4002, Vienna
- Brazil (7):
  - Hospital Sao Rafael Instituto D'Or da Bahia Site Number : 7608, Salvador, Estado de Bahia
  - Uniao Oeste Paranaense de Estudos e Combates ao Cancer Site Number : 7610, Cascavel, Paraná
  - Hospital De Clinicas De Porto Alegre Site Number : 7605, Porto Alegre, Rio Grande do Sul
  - Hospital Santa Marcelina Site Number : 7611, São Paulo, São Paulo
  - CEMEC Oncologica do Brasil Site Number : 7606, Belém
  - HEMORIO - Instituto Estadual de Hematologia Arthur de Siqueira Cavalcanti Site Number : 7609, Rio de Janeiro
  - Hospital do Servidor Publico Estadual de Sao Paulo Site Number : 7607, São Paulo
- Canada (3):
  - Investigational Site Number : 12404, Edmonton, Alberta
  - Investigational Site Number : 12406, Toronto, Ontario
  - CHU Sainte-Justine_Investigational site number 12405, Montreal, Quebec
- Chile (3):
  - Investigational Site Number : 15201, La Serena, Coquimbo Region
  - Investigational Site Number : 15204, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 15202, Viña del Mar, Región de Valparaíso
- China (12):
  - Wuhan Union Hospital of Tongji Medical College of HUST - Investigational Site Number: 15601, Wuhan, Hubei
  - Shengjing Hospital of China Medical University - Investigational Site Number: 15603, Shenyang, Liaoning
  - Shaanxi Provincial People's Hospital - Investigational Site Number: 15607, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University - Investigational Site Number: 15605, Jinan, Shandong
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences - Investigational Site Number: 15602, Tianjin, Tianjin Municipality
  - Second Affiliated Hospital of Kunming Medical University - Investigational Site Number: 15604, Kunming, Yunnan
  - Investigational Site Number : 15611, Hangzhou
  - Investigational Site Number : 15608, Hefei
  - Investigational Site Number : 15610, Nanchang
  - Investigational Site Number : 15613, Tangshan
  - Investigational Site Number : 15609, Wuxi
  - Investigational Site Number : 15614, Zhenjiang
- France (7):
  - Investigational Site Number : 25014, Angers
  - Investigational Site Number : 25011, Créteil
  - Investigational Site Number : 25010, Dijon
  - Investigational Site Number : 25009, Nantes
  - Investigational Site Number : 25008, Paris
  - Investigational Site Number : 25012, Paris
  - Investigational Site Number : 25007, Pessac
- Germany (4):
  - Investigational Site Number : 27610, Berlin
  - Investigational Site Number 27612, Düsseldorf
  - Investigational Site Number : 27613, Frankfurt am Main
  - Investigational Site Number : 27611, Recklinghausen
- Hungary (5):
  - Investigational Site Number : 34803, Budapest
  - Investigational Site Number : 34805, Debrecen
  - Investigational Site Number : 34801, Győr
  - Investigational Site Number : 34804, Nyíregyháza
  - Investigational Site Number : 34802, Székesfehérvár
- Israel (5):
  - Investigational Site Number : 37605, Haifa
  - Investigational Site Number : 37606, Kfar Saba
  - Investigational Site Number : 37607, Tel Aviv
  - Investigational Site Number : 37608, Tel Litwinsky
  - Investigational Site Number : 37609, Ẕerifin
- Italy (6):
  - Investigational Site Number : 38014, Florence, Tuscany
  - Investigational Site Number : 38012, Bologna
  - Investigational Site Number : 38015, Milan
  - Investigational Site Number : 38013, Milan
  - Investigational Site Number : 38010, Trieste
  - Investigational Site Number : 38011, Vicenza
- Japan (12):
  - Investigational Site Number : 39214, Tsuchiura-shi, Ibaraki
  - Investigational Site Number : 39205, Kanazawa, Ishikawa-ken
  - Investigational Site Number : 39207, Sagamihara-shi, Kanagawa
  - Investigational Site Number : 39202, Suita-shi, Osaka
  - Investigational Site Number : 39201, Iruma-gun, Saitama
  - Investigational Site Number : 39208, Bunkyo-ku, Tokyo
  - Investigational Site Number : 39210, Meguro-ku, Tokyo
  - Investigational Site Number : 39204, Setagaya City, Tokyo
  - Investigational Site Number : 39209, Sumida-ku, Tokyo
  - Investigational Site Number : 39212, Chiba
  - Investigational Site Number : 39203, Hiroshima
  - Investigational Site Number : 39206, Saitama-shi
- Mexico (6):
  - Investigational Site Number : 48401, Monterrey, Nuevo León
  - Investigational Site Number : 48402, Chihuahua City
  - Investigational Site Number : 48405, Delegacion Benito Juarez
  - Investigational Site Number : 48404, Durango
  - Investigational Site Number : 48406, Mexico City
  - Investigational Site Number : 48403, Zapopan
- Erasmus MC_Investigational Site Number 52801, Rotterdam, Netherlands
- Norway (2):
  - Investigational Site Number : 57802, Bergen
  - Investigational Site Number : 57801, Grålum
- Poland (6):
  - Investigational Site Number : 61617, Piła, Greater Poland Voivodeship
  - Investigational Site Number : 61609, Słupsk, Pomeranian Voivodeship
  - Investigational Site Number : 61615, Gdynia
  - Investigational Site Number : 61614, Poznan
  - Investigational Site Number : 61612, Warsaw
  - Investigational Site Number : 61613, Wroclaw
- Russia (7):
  - Investigational Site Number : 64307, Moscow
  - Investigational Site Number : 64305, Moscow
  - Investigational Site Number : 64304, Novosibirsk
  - Investigational Site Number : 64301, Pyatigorsk
  - Investigational Site Number : 64302, Saint Petersburg
  - Investigational Site Number : 64306, Samara
  - Investigational Site Number : 64303, Tula
- Singapore (3):
  - Investigational Site Number : 70201, Singapore
  - Investigational Site Number : 70202, Singapore
  - Investigational Site Number : 70203, Singapore
- South Korea (5):
  - Investigational Site Number : 41004, Busan, Busan
  - Investigational Site Number : 41001, Suwon, Gyeonggi-do
  - Investigational Site Number : 41003, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 41005, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number : 41006, Seoul, Seoul-teukbyeolsi
- Spain (9):
  - Investigational Site Number : 72408, Málaga, Málaga
  - Investigational Site Number : 72407, Valencia, Valenciana, Comunidad
  - Investigational Site Number : 72412, Barcelona
  - Investigational Site Number : 72414, Barcelona
  - Investigational Site Number : 72409, Barcelona
  - Investigational Site Number : 72416, Burgos
  - Investigational Site Number : 72410, Madrid
  - Investigational Site Number : 72411, Murcia
  - Investigational Site Number : 72413, Seville
- Thailand (5):
  - Investigational Site Number : 76405, Bangkok
  - Investigational Site Number : 76404, Bangkok
  - Investigational Site Number : 76402, Chiang Mai
  - Investigational Site Number : 76401, Khon Kaen
  - Investigational Site Number : 76403, Songkhla
- Turkey (Türkiye) (4):
  - Investigational Site Number 79208, Ankara
  - Investigational Site Number 79210, Istanbul
  - Investigational Site Number 79206, Izmir
  - Investigational Site Number 79209, Kayseri
- Ukraine (3):
  - Investigational Site Number : 80408, Dnipropetrovsk
  - Investigational Site Number : 80409, Kryvyi Rih
  - Investigational Site Number : 80410, Kyiv
- United Kingdom (7):
  - Investigational Site Number : 82607, London, London, City of
  - Investigational Site Number : 82604, Harrow
  - Investigational Site Number : 82606, London
  - Investigational Site Number : 82609, London
  - Investigational Site Number : 82603, Manchester
  - Investigational Site Number : 82605, Norfolk
  - Investigational Site Number : 82608, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Kuter DJ, Ghanima W, Cooper N, Liebman HA, Zhang L, Hu Y, Miyakawa Y, Homenda W, Galindo LEM, Basquiera AL, Tan CW, Saydam G, Hutter-Kronke ML, Chai-Adisaksopha C, Gomez-Almaguer D, Tran H, Shin HJ, Dantas da Cunha Junior A, Lazar Z, Izquierdo CP, Kirgner I, Lucchini E, Kuzmina G, Fillitz M, Audia S, Taparia M, Cordoba M, Diab R, Yao M, Gouia I, Lee M, Daak A. Safety and efficacy of rilzabrutinib vs placebo in adults with immune thrombocytopenia: the phase 3 LUNA3 study. Blood. 2025 Jun 12;145(24):2914-2926. doi: 10.1182/blood.2024027336. PMID 40090011
- [Derived] Lin J, Radhakrishnan J. What Are Baskets, Umbrellas, and Platforms Doing in Nephrology Clinical Trials? J Am Soc Nephrol. 2025 Feb 3;36(8):1652-1654. doi: 10.1681/ASN.0000000648. No abstract available. PMID 39899371
- [Derived] Kuter DJ, Bussel JB, Ghanima W, Cooper N, Gernsheimer T, Lambert MP, Liebman HA, Tarantino MD, Lee M, Guo H, Daak A. Rilzabrutinib versus placebo in adults and adolescents with persistent or chronic immune thrombocytopenia: LUNA 3 phase III study. Ther Adv Hematol. 2023 Oct 18;14:20406207231205431. doi: 10.1177/20406207231205431. eCollection 2023. PMID 37869360